CLINICAL TRIAL: NCT03178201
Title: Study of the Phosphoinositide-3-Kinase-Delta Inhibitor TGR-1202 in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: TGR1202 in Relapsed and Refractory Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR1223
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Follicular Lymphoma
Keywords: Relapsed follicular lymphoma; Refractory follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — umbralisib; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TGR-1202 (Experimental): Patients with relapsed or refractory grade 1, 2, or 3A follicular lymphoma will receive TGR-1202.
  Interventions: Drug: TGR-1202

INTERVENTIONS:
Drug: TGR-1202 — Treatment will be self-administered on an outpatient basis. Patients will take TGR-1202 800 mg, oral, one tablet daily on a continuous basis. Each cycle lasts 28 days.
  Other Names: formerly as RP5307

SUMMARY:
The primary objective is to determine the overall response rate (ORR) of TGR-1202 in R/R FL.

Secondary Objectives

* Determine the genetic and other novel biological markers that may be predictive of response or resistance to TGR-1202 in patients with relapsed or refractory FL.
* Describe the Progression Free Survival (PFS), Duration of Response (DoR) after treatment with TGR-1202.
* Describe the number of dose delays and dose reductions and other safety profile.

DETAILED DESCRIPTION:
This is an open label, phase II study of TGR-1202 in patients with relapsed or refractory (R/R) Grade 1, 2, or 3A follicular lymphoma (FL). FL is the most common subtype of indolent lymphoma. The prognosis of FL depends on the histologic grade, stage, treatment and age of the patient. More recently, efforts have been made to find novel regimens for the treatment of relapsed FL that do not contain non-specific cytotoxic agents.

One of the important goals of this phase II study is to discover novel genetic, biochemical, and immunological markers that are associated with the response and safety of TGR-1202 in patients with FL. TGR-1202 blocks PI3K, a signal that is required for cancer to grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of grade 1, 2, or 3A FL.
* Relapse following first line immunotherapy or chemoimmunotherapy. There is no upper limit to the number of therapies received prior to study entry. Prior therapies may include high-dose therapy with autologous stem cell rescue.
* Measurable Disease according to the Lugano classification.
* Lymphoma that is amenable to safe pre-treatment and post-treatment biopsy. The safety of the procedures will be determined by the treating physician and the surgeon in consultation with the PI, and in accordance with standard clinical practice. Acceptable sites of disease include, for example: (1) palpable tumor mass that is accessible under direct visualization or sonogram, (2) non-palpable tumor tissue that is accessible for biopsy under computed tomography (CT) or sonogram guidance, (3) bone marrow.
* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patients must have adequate organ and marrow function as defined below:

  1. absolute neutrophil count >1,000/microliter
  2. platelet count ≥50,000/microliter
  3. bilirubin <1.5 x institutional upper limit of normal
  4. aspartate transaminase (AST, SGOT)/alanine transaminase (ALT, SGPT) <3.0 x institutional upper limit of normal
  5. Serum creatinine <2.0 x institutional upper limit of normal or creatinine clearance >50 mL/min (according to the Cockcroft and Gault equation).
* Negative serum pregnancy test within 7 days prior to Cycle 1/Day 1 for women of childbearing potential.
* All women of childbearing potential must agree to use an effective barrier method of contraception, as described in Appendix 4, during the treatment period and for at least 1 month after discontinuation of the study drug. Male subjects should use effective barrier method of contraception during the treatment period and for at least 1 month after discontinuation of the study drug
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Grade 3B FL or evidence of transformation to a more aggressive lymphoma
* Prior and concomitant therapy:

  1. Prior exposure to any PI3 Kinase inhibitor
  2. Exposure to chemotherapy, radiotherapy, or immunotherapy within 3 weeks prior to entering the study or lack of recovery from adverse events (AE) due to previously administered treatments.
  3. Ongoing chronic immunosuppressants (e.g. cyclosporine) or systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone prior to the start of the study drug.
  4. Other concurrent investigational agents during the study period.
* Prior allogeneic stem cell transplant
* Central nervous system lymphoma, including lymphomatous meningitis
* Acute intercurrent illness including, but not limited to, active infection, unstable congestive heart failure, unstable angina pectoris, psychiatric illness or any social situation that would limit compliance with study participation requirements in the judgement of the investigator.
* Major surgery performed within 4 weeks of study entry
* Pregnant or nursing women
* Active concurrent malignancy (except non-invasive non-melanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasia). If there is a history of prior malignancy, the patient must be disease-free for ≥ 3-years at the time of study entry.
* Documented Human Immunodeficiency Virus (HIV)-infection
* Active hepatitis A, hepatitis B, or hepatitis C infection
* History of tuberculosis treatment within 2 years of study entry
* Administration of a live vaccine within 6 weeks of first dose of study drug
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy)
* Lymphoma that is not amenable for mandatory pre- and post-treatment biopsy as described in the inclusion criteria.
* Unstable or severe uncontrolled medical condition (e.g. unstable cardiac function, unstable pulmonary condition, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the patient associated with his or her participation in the study
* Clinically significant cardiovascular abnormalities such as:

  1. QTc ≥ 470 msec.
  2. Angina not well-controlled by medication
  3. Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac/vascular stenting within 6 months of enrollment
  4. Symptomatic or documented congestive heart failure that meets New York Heart Association (NYHA) Class III to IV definitions;
  5. History of stroke within the last 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Changchun Deng, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TGR-1202
Started | 5
Completed | 0
Not Completed | 5
Not completed — Off study | 5

BASELINE CHARACTERISTICS:
Arm/Group | TGR-1202
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The sum of patients with partial responses and complete responses.
Time Frame: Up to 3 years
Population: The data was not collected or analyzed due to the study was terminated prematurely due to slow to accrual and PI left the institution.
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS) After Treatment With TGR-1202
Description: The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DoR) After Treatment With TGR-1202
Description: The time of initial response until documented tumor progression.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Dose Delays
Description: The number of instances of patients having a dose of study drug delayed 1 or more days.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Dose Reductions
Description: The number of instances of patients having to reduce the dosage of study drug based on specified toxicities.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] broken down by adverse event and CTCAE v4.0 grade of each event.
Time Frame: Up to 3 years
Population: as for outcome 1
Arm/Group | TGR-1202
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year post treatment
Arm/Group | TGR-1202
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03178201/Prot_SAP_000.pdf